CLINICAL TRIAL: NCT02400151
Title: Vascular and Metabolic Effects of Vitamin D Supplementation Associated With Lifestyle Management in Obese Adolescents: Prospective, Randomized, Controlled Trial
Brief Title: Vascular and Metabolic Effects of Vitamin D Supplementation Associated With Lifestyle Management in Obese Adolescents
Acronym: VIDADO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: UMR1260 NORT Nutrition, Obésité et Risque Thrombotique (Unknown); EA4278 PEC Laboratoire de Pharm-Ecologie Cardiovasculaire (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LOCAL/2015/APM-01; 2015-000060-34 (EudraCT Number)
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2017-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Non-Obese group (Other): Non-obese patients will be recruited and frequency matched to obese groups according to sex and level of sexual maturation.
  Intervention: Normal control
  Interventions: Other: Normal control
- Obese group, Vitamin D (Experimental): Subjects randomized to this group will receive vitamin D supplementation. They are recruited from the St Pierre Institute at Palavas-les-Flots, France.
  Intervention: 3 months lifestyle and dietary management Intervention: Vitamin D supplementation
  Interventions: Drug: Vitamin D supplementation; Other: 3 months lifestyle and dietary management
- Obese group, placebo (Placebo Comparator): Subjects randomized to this group will receive a placebo supplement. They are recruited from the St Pierre Institute at Palavas-les-Flots, France.
  Intervention: 3 months lifestyle and dietary management Intervention: Placebo
  Interventions: Drug: Placebo; Other: 3 months lifestyle and dietary management

INTERVENTIONS:
Drug: Vitamin D supplementation — Patients randomized to this group will receive 4000 UI of Vitamin D3 per day for 90 days.
  Arms: Obese group, Vitamin D
Drug: Placebo — Patients randomized to this group will receive placebo for 90 days.
  Arms: Obese group, placebo
Other: 3 months lifestyle and dietary management — Lifestyle and dietary management at the Saint Pierre Institute (Palavas-les-Flots, France) occurs for three months. Nutritionally speaking, each child or adolescent receives a controlled and balanced diet, consistent with the recommendations appropriate for his/her age, slightly hypocaloric or normocaloric. This dietary approach is complemented by a nutrition education program and supervision by a doctor and a dietician. Three hours of exercise training per week are scheduled; these sessions include adapted aerobic activities supervised by instructors and educators at the center.
  Arms: Obese group, Vitamin D; Obese group, placebo
Other: Normal control — Patients in this group do not have experimental intervention in order to provide measures of a real-life control group.
  Arms: Non-Obese group

SUMMARY:
The main objective of this study is to analyze in a population of obese adolescents, the effect of vitamin D3 supplementation in addition to lifestyle and dietary management on vascular function assessed by the change between M0 and M3 of endothelium-dependent vasorelaxation measured at the brachial artery (Flow-Mediated Dilation).

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. To analyze in obese adolescents, the effect of the addition of vitamin D3 supplementation on metabolic and vascular function.

B. To compare the relationships between food intake, metabolic, inflammatory, oxidative stress and vitamin D status, and vascular dysfunction between obese and normal weight subjects.

C. To evaluate the effects of sun exposure variations on relationships described in Objective B by comparing the observed parameters at baseline and at the end of the three month follow-up period, in non-supplemented obese adolescents and adolescents of normal weight.

D. To identify biomarkers (metabolic signatures) in obese adolescents associated with vitamin D deficiency and vascular function.

E. To evaluate in obese adolescents, the effects of vitamin D supplementation on the metabolome (metabolic signature).

F. To evaluate the effects of lifestyle and dietary management on these biomarkers (in the "control group").

For these targets (A to F), all teenagers will be classified according to three levels of skin pigmentation.

G. Establish a biobank of samples taken at baseline and at 3 months.

ELIGIBILITY:
General Inclusion Criteria:

* The patient's legal representatives must have given their informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Sexual maturation of at least Tanner stage 2

Inclusion criteria for the patient population

* The subject has a body mass index corresponding to grade 2 obesity according to the curves described by Rolland-Cachera et al (1991)
* Absence of at least 5% of total weight over the last 3 months

Inclusion criteria for the control population

* The subject has a body mass index < 90th percentile

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection
* The patient's legal representative(s) refuse(s) to sign the consent
* It is impossible to correctly inform the patient or his/her legal representative(s)
* The patient has a contraindication for physical activity (joint, heart or other)
* The subject does at least 3 hours of extracurricular physical activity per week
* The subject has a concomitant illness, a history of first-degree cardiovascular disease, abnormal glucose tolerance (pre-diabetes or diabetes).
* Active smoking
* Known dyslipidemia (particularly hypercholesterolemia).
* The subject regularly takes food and vitamin supplements and refuses to stop taking these during the study (in case of disruption of these supplements, a wash-out stopping period of 3 weeks is required).
* BMI corresponding to a grade 1 obesity according to the Rolland-Cachera et al. (1991) curves.
* Secondary or known genetic obesity.
* Known hypersensitivity to vitamin D.
* Hypercalcemia, hypercalciuria, calcium lithiasis

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2016-07-04 (Actual); Study Completion 2016-07-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Flow Mediated Dilation (%) at the brachial artery | 3 months

SECONDARY OUTCOMES:
Change from baseline in Nitrate Mediated Dilation (%) at the brachial artery | 3 months
Change from baseline in carotid compliance (mm^2mmHg^-1) | 3 months
Change from baseline in brachial compliance (mm^2mmHg^-1) | 3 months
Change from baseline in arterial wave speed (m*s^-1) | 3 months
Usual Vitamin D intake according to food questionnaire | Baseline
Change from baseline in blood 25(OH)D levels (mmol*L^-1) | 3 months
Change from baseline in blood parathyroid hormone levels (mmol*L^-1) | 3 months
Change from baseline in serum calcium levels (mmol*L^-1) | 3 months
Change from baseline in blood total protein levels (g*L^-1) | 3 months
Change from baseline in Homeostatic model assessment Insulin Resistance | 3 months
Change from baseline in the ratio Low Density Lipoprotein/High Density Lipoprotein | 3 months
Change from baseline in Triglyceride levels | 3 months
Change from baseline in Acetylcholine-Cutaneous Blood Flow peak | 3 months
Change from baseline in Sodium nitroprussiate-Cutaneous Blood Flow peak (%) | 3 months
Change from baseline in Insulin-Cutaneous Blood Flow peak (%) | 3 months
Change from baseline in TNF-alpha (pg*mL^-1) | 3 months
Change from baseline in IL-6 (pg*mL^-1) | 3 months
Change from baseline in High sensitivity C-reactive protein (pg*mL^-1) | 3 months
Change from baseline in leptin (pg*mL^-1) | 3 months
Change from baseline in adiponectin (pg*mL^-1) | 3 months
Change from baseline in SuperOxyde Dismutase (U*gHb^-1) | 3 months
Change from baseline in Isoprostanes (ng*L^-1) | 3 months
Change from baseline in nitrite-nitrate (µmol*L^-1) | 3 months
Change from baseline in PAI-1 (µmol*L^-1) | 3 months
Metabolomic profile | baseline
Metabolomic profile | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Perez Martin, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - Institut Saint Pierre, Palavas-les-Flots

REFERENCES:
- [Result] Vinet A, Morrissey C, Perez-Martin A, Goncalves A, Raverdy C, Masson D, Gayrard S, Carrere M, Landrier JF, Amiot MJ. Effect of vitamin D supplementation on microvascular reactivity in obese adolescents: A randomized controlled trial. Nutr Metab Cardiovasc Dis. 2021 Jul 22;31(8):2474-2483. doi: 10.1016/j.numecd.2021.04.025. Epub 2021 May 10. PMID 34090775